CLINICAL TRIAL: NCT02942394
Title: Non-interventional, Multicenter, Multinational Venous Stent Study for the Treatment of the Post-thrombotic Syndrome With Common Iliac Vein Compression
Brief Title: Treatment of the Postthrombotic Syndrome With the Oblique Stent - TOPOS Study
Status: Completed | Type: Observational
Sponsor: Optimed Medizinische Instrumente GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: SONIS15473
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Post-thrombotic Syndrome; Iliac Vein Compression Syndrome
MeSH Terms: conditions — Postthrombotic Syndrome; May-Thurner Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: sinus-Obliquus Stent System

SUMMARY:
Primary objective:

To assess the efficacy of the stents (sinus-Obliquus stent for the common iliac vein, the sinus-XL Flex stent or sinus-Venous stent for the external iliac and common femoral veins) by evaluating different gradations of patency rates, patient's rating of disease severity and quality of life in patients with post-thrombotic syndrome and concomitant common iliac vein compression.

Secondary objective:

To assess long-term safety of venous stenting

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged ≥18 years
2. Post-thrombotic syndrome (Villalta score >4 points) due to iliac vein thrombosis with or without femoral deep vein thrombosis
3. Evidence of venous stenosis in common iliac vein >50% confirmed by venography (CT or MRI) or intravascular ultrasound (IVUS)
4. Use of sinus-Obliquus stent for unilateral common iliac vein stenosis
5. If stent extension is required either sinus-XL Flex or sinus-Venous stents must have been used for stenoses >50% confirmed by venography (CT or MRI) or IVUS in external iliac and common femoral veins

Exclusion Criteria:

1. Pregnancy, breast-feeding or birth-giving during the last 30 days
2. Life expectancy <6 months
3. Iliofemoral DVT less than 3 months ago
4. Permanently immobile patient (wheelchair user or bed-ridden patient)
5. Allergy to Nitinol
6. Patient's target vessel(s) has/have been stented before
7. Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible impact of the study
8. Patients in custody by juridical or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with post-thrombotic syndrome and concomitant common iliac vein compression.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-12; Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Primary Patency Rate | After 3 months up to a follow-up of 2 years.

SECONDARY OUTCOMES:
Primary Assisted Patency Rate | After 3 months up to a follow-up of 2 years.
Secondary Patency Rate | After 3 months up to a follow-up of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof. Dr. med., Principal Investigator — Director Clinic for Angiology Universitätsspital Zürich
Locations (7):
- Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- Germany (3):
  - Karolinen Hospital Arnsberg, Arnsberg
  - Medizinische Universitätsklinik Heidelberg, Heidelberg
  - Universität des Saarlandes, Homburg
- Maastricht University Hospital MUMC+, Maastricht, Netherlands
- Switzerland (2):
  - INSELSPITAL, Universitätsspital Bern, Bern
  - Universitätsspital Zürich, Zurich